CLINICAL TRIAL: NCT04000399
Title: BRITEPath, Component 3 of iCHART (Integrated Care to Help At-Risk Teens)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephanie Stepp, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Study18120080; P50MH115838-02 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Ultimately, this study design was an open trial after unsuccessful attempts to maintain initial recruitment sites in the study.
  This study initially attempted to use a stepped wedge design, which involves the sequential random rollout of an intervention over 2 time periods. Following a baseline period in which no clusters (= practices) are exposed to the intervention, the crossover is typically in one direction, from control to intervention and continues until both of the clusters have crossed-over to receive the intervention, with observations taken from each cluster and at each time period.
Masking Description: Outcomes assessors will be masked to the intervention condition at follow-up assessment timepoints.
  See notes on pre-assignment details in participant flow related to study model single arm vs. multi arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRITEPath (Experimental): Participants will receive the components in BRITEPath from a mental health (MH) clinician trained by the study staff/PI's on how to implement BRITE safety planning with fidelity.
  First, the MH clinician will review possible barriers to implementation of the safety plan and problem-solve appropriately with patient and parent(s); (2) BRITE is the emotion regulation/safety planning app loaded on the patient's smartphone that populated with support from Guide2BRITE.; and (3) BRITEBoard, a clinician dashboard that shows app use, change in distress and symptoms ratings, and can be used for shared decision making with parents, patients, and PCPs. Clinicians will review adolescent's skill development and app content with parents. Prior to discharge or following acute increases in suicide risk.
  Interventions: Behavioral: BRITEPath

INTERVENTIONS:
Behavioral: BRITEPath — BRITEPath will guide co-located mental health clinicians in the use of an emotion regulation and safety planning app (BRITE) to be loaded on the phone of depressed and suicidal adolescents in order to improve depression and reduce the likelihood of a suicide attempt.

SUMMARY:
BRITEPath (BP) aims to support co-located mental health clinicians in the development of a high quality, effective, and personalized safety plan for referred patients who screen positive for depression and/or suicidal ideation.

BRITEPath utilizes BRITE, a safety planning and emotion regulation app that is loaded on the patient's smart phone and has previously been shown to be well accepted and to reduce suicide attempts compared to usual care in psychiatric inpatients (HR = 0.49). To support mental health clinicians in the development of effective safety plans, study investigators will develop Guide2Brite (G2B), which provides step-by-step instructions for the mental health clinician on how to populate BRITE onto the patient's smartphone and BRITEBoard, a clinician dashboard that tracks patient symptoms, app use, and rating on helpfulness of different interventions assessed through BRITE.

DETAILED DESCRIPTION:
Delivery of Interventions:

BRITEPath has 3 components:1) BRITE, an emotion regulation and safety planning phone app that is delivered by a co-located mental health (MH) clinician to adolescents at the time of their first therapy appointment; 2) Guide2Brite, which will guide the co-located MH clinician in working with the adolescent to population content onto BRITE; and 3) BRITEBoard, which is a clinician dashboard delivered to the MH clinician and PCP.

Assignment of Interventions:

This study utilized an open trial design. A stepped wedge design was originally proposed and efforts were made to adhere to this study design, however after a year of low recruitment and resultant recruitment sites pulling out the of the study, the overall study design was changed to an open trial. Additional recruitment sites were onboarded to the study and provided with the intervention arm in order to obtain feasibility data on the intervention components of the study. As a result of the change, there are some TAU participants included in this study. For reference a stepped wedge design involves the sequential random rollout of an intervention over two time periods. Following a baseline period in which no clusters (=practices) are exposed to the intervention, the crossover is typically in one direction, from control to intervention and continues until both of the clusters have crossed-over to receive the intervention, with observations taken from each cluster and at each time period.

Study investigators will pilot BRITEPath in community pediatric and mental health practices using a stepped wedge design (n =50 adolescents).

Hypothesis: The use of BRITEPath will decrease depressive symptoms, distress, and suicidality (any self-injurious ideation, urges, or behavior) as well as improve overall functioning compared to TAU.

Of note: Study investigators initially intended to do a cost analysis as a secondary outcome measure, but it was later decided that the analysis will not be done in this pilot phase of testing and will instead be completed during the Phase 2 RCT.

ELIGIBILITY:
Inclusion Criteria:

* Youth aged 12-26 yo
* Own a device (e.g. smartphone, ipod, tablet) with capability to download BRITE app
* Biological or adoptive parent is willing to provide informed consent for teen to participate
* Youth speaks and understands English
* Positive PHQ score or provider determines youth has depressive symptoms based on clinical interaction and refers youth to the study (in cases when PHQ is not available and study staff will complete the PHQ during the screening) OR Provider can refer if they are unclear if symptoms are depressive and PHQ scoring will be used to determine youth's eligibility. OR Screening Wizard screening questionnaire (which includes the PHQ and depressive symptom questions) indicates depression OR provider/parent have concern that youth/patient has a mood or behavioral problem
* Family agrees to see an (embedded) MH therapist at the practice

PHQ scores:

Score of 8 or higher on PHQ-8 -or- Score of 1 or higher on #9 of PHQ-9 suicidality item

Exclusion Criteria:

Non English speaking No parent willing to provide informed consent No cell phone capability of downloading BRITE app Is currently experiencing mania or psychosis Evidence of an intellectual or developmental disorder (IDD) Life threatening medical condition that requires immediate treatment (included emergent suicidality, homicidality, abuse/neglect, or other mental or physical condition) Other cognitive or medical condition preventing youth from understanding study and/or participating.

Currently receiving MH treatment/currently satisfied with treatment

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Stepp, PhD, Principal Investigator — University of Pittsburgh; David Brent, MD, Study Director — University of Pittsburgh
Locations (6):
- United States (6):
  - Northwell Hospital, Hyde Park, New York
  - Children's Community Pediatrics (CCP-Moon) of Children's Hospital of Pittsburgh of UPMC, Moon Township, Pennsylvania
  - STAR-Center, Pittsburgh, Pennsylvania
  - Wesley Family Services, Pittsburgh, Pennsylvania
  - Children's Community Pediatrics (CCP-Wexford) of Children's Hospital of Pittsburgh of UPMC, Wexford, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication.
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants were assigned to the single arm/group originally specified in the protocol and started Treatment as Usual but, due to a protocol amendment, these participants were not crossed over, and all subsequent participants were assigned to the BritePath intervention only. Thus we consider this a single arm study.
Groups:
- BritePath: Participants will receive the components in BRITEPath from a mental health (MH) clinician trained by the study staff/PI's on how to implement BRITE safety planning with fidelity.
  First, the MH clinician will review possible barriers to implementation of the safety plan and problem-solve appropriately with patient and parent(s); (2) BRITE is the emotion regulation/safety planning app loaded on the patient's smartphone that populated with support from Guide2BRITE.; and (3) BRITEBoard, a clinician dashboard that shows app use, change in distress and symptoms ratings, and can be used for shared decision making with parents, patients, and PCPs. Clinicians will review adolescent's skill development and app content with parents. Prior to discharge or following acute increases in suicide risk.
  BRITEPath: BRITEPath will guide co-located mental health clinicians in the use of an emotion regulation and safety planning app (BRITE) to be loaded on the phone of depressed and suicidal adolescents in order to improve depression and reduce the likelihood of a suicide attempt.
- Treatment As Usual (TAU): Participants in the TAU group will not receive the Brite emotion regulation/safety planning app. If participants in the TAU group are determined to be at risk for suicidal ideation or behavior, usual care of a paper-based safety plan will be utilized.
Period: Overall Study
Arm/Group | BritePath | Treatment As Usual (TAU)
Started | 38 | 5
Completed | 38 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: 3 participants were recruited, completed the consenting process (where we collect age data), and were randomized, but did not complete the baseline or follow up visits where the rest of our demographic information is collected. These 3 pts also engaged in use of the app/intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | BritePath | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 38 | 5 | 43
Age, Categorical [Count of Participants; unit: Participants] — Measure Analysis Population Description: 3 participants were recruited, completed the consenting process (where we collect age data), and were randomized, but did not complete the baseline or follow up visits where the rest of our demographic information is collected. These 3 pts also engaged in use of the app/intervention.
  Participants
    <=18 years | 31 | 5 | 36
    Between 18 and 65 years | 7 | 0 | 7
    >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: 3 participants were recruited, completed the consenting process (where we collect age data), and were randomized, but did not complete the baseline visit where the rest of our demographic information is collected.
  Participants
    Male: number analyzed (Participants) | 35 | 5 | 40
    Male | 8 | 1 | 9
    Female: number analyzed (Participants) | 35 | 5 | 40
    Female | 26 | 4 | 30
    Non-binary/ Queer: number analyzed (Participants) | 35 | 5 | 40
    Non-binary/ Queer | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 participants were recruited, completed the consenting process (where we collect age data), and were randomized, but did not complete the baseline visit where the rest of our demographic information is collected.
  Participants
    number analyzed (Participants) | 35 | 5 | 40
    Hispanic or Latino | 7 | 0 | 7
    Not Hispanic or Latino | 28 | 5 | 33
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 participants were recruited, completed the consenting process (where we collect age data), and were randomized, but did not complete the baseline visit where the rest of our demographic information is collected.
  Participants
    number analyzed (Participants) | 35 | 5 | 40
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 1 | 0 | 1
    White | 25 | 4 | 29
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 38 | 5 | 43

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity
Description: Total scores from the Patient Health Questionnaire (PHQ-9) will be used to assess depression severity, as a primary outcome. The PHQ-9 is 9 items with scoring ranging from 0-27. The higher the score, the more severe the depression symptoms are. A score of 0-4=no depression; 5-9=mild depression; 10-14=moderate depression; 15-19=moderately severe depression; 20-27=severe depression symptoms.
Time Frame: At Baseline phone visit
Population: 3 participants did not complete baseline or follow up visits. These 3 individuals completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 35 | 5
score on a scale | 12.9 (4.8) | 9.2 (5.8)

2. Primary Outcome: Depression Severity
Description: as for outcome 1
Time Frame: At 4 week follow up after Baseline
Population: Of the 38 participants assigned to BRITEPath, 32 completed the PHQ-9 at the 4 week follow-up timepoint. Of the 5 participants assigned to TAU, 4 completed the PHQ-9 at the 4 week follow-up timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 32 | 4
score on a scale | 10.9 (6) | 5.5 (1.3)

3. Primary Outcome: Depression Severity
Description: as for outcome 1
Time Frame: At 12 week follow up after Baseline
Population: Of the 38 participants assigned to BRITEPath, 32 completed the PHQ-9 at the 12 week follow-up timepoint. Of the 5 participants assigned to TAU, 4 completed the PHQ-9 at the 12 week follow-up timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 32 | 4
score on a scale | 10.4 (5.4) | 9.5 (1.7)

4. Primary Outcome: Suicidal Ideation and Behavior
Description: Suicidal attempt & ideation will be measured through the Columbia Suicide Severity Rating Scale (C-SSRS) and the Patient Health Questionnaire (PHQ-9). Assign score of 0 if no ideation/behavior present and assign a score of 1 if ideation/behavior present. A "yes" answer any time during treatment to question 9 on the PHQ-9 indicates suicidal ideation. A "yes" answer any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 7-10) on the C-SSRS. C-SSRS Categories 7-10 are as follows: 7-Aborted Attempt 8-Interrupted Attempt 9-Actual Attempt (non-fatal) 10-Completed Suicide. Any score greater than 0 is important/may indicate need for intervention.
Time Frame: At Baseline phone visit
Population: Of the 38 participants in BRITEPath intervention, only 35 completed CSSRS. All 5 from TAU completed CSSRS.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 35 | 5
score on a scale
  PHQ-9 Question 9 (ideation) | 1.1 (1) | 0 (0)
  C-SSRS Category 7: Aborted Attempt | 0.1 (0.2) | 0 (0)
  C-SSRS Category 8: Interrupted Attempt | 0 (0) | 0 (0)
  C-SSRS Category 9: Actual Attempt (non-fatal) | 0.1 (0.3) | 0 (0)
  C-SSRS Category 10: Completed Suicide | 0 (0) | 0 (0)

5. Primary Outcome: Suicidal Ideation and Behavior
Description: as for outcome 4
Time Frame: At 4 week follow up after Baseline
Population: Of the 38 participants assigned to BRITEPath, 32 completed the C-SSRS at the 4 week follow-up timepoint. Of the 5 participants assigned to TAU, 4 completed the C-SSRS at the 4 week follow-up timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 32 | 4
score on a scale
  PHQ-9 Question 9 (ideation) | 0.9 (1) | 0 (0)
  C-SSRS Category 7: Aborted Attempts | 0 (0) | 0 (0)
  C-SSRS Category 8: Interrupted Attempts | 0 (0.2) | 0 (0)
  C-SSRS Category 9: Actual Attempts (non-lethal) | 0.1 (0.2) | 0 (0)
  C-SSRS Category 10: Completed Suicide | 0 (0) | 0 (0)

6. Primary Outcome: Suicidal Ideation and Behavior
Description: as for outcome 4
Time Frame: At 12 week follow up after Baseline
Population: Of the 38 participants assigned to BRITEPath, 32 completed the C-SSRS at the 12 week follow-up timepoint. Of the 5 participants assigned to TAU, 4 completed the C-SSRS at the 12 week follow-up timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 32 | 4
score on a scale
  PHQ-9 Question 9 (ideation) | 0.6 (0.8) | 0 (0)
  C-SSRS Category 7: Aborted Attempts | 0 (0) | 0 (0)
  C-SSRS Category 8: Interrupted Attempts | 0.1 (0.2) | 0 (0)
  C-SSRS Category 9: Actual Attempts (non-lethal) | 0 (0) | 0 (0)
  C-SSRS Category 10: Completed Suicide | 0 (0) | 0 (0)

7. Primary Outcome: Quality of Life and Social/Emotional Functioning
Description: The Pediatric Quality of Life Inventory Version 4.0 (PedsQOL) will be used to assess overall quality of life and functioning, as a primary outcome. The PEDSQOL has 23 items and ranges in score from 0-92. It is broken down into 4 subdomains of physical functioning, emotional functioning, social functioning, and work/school (psychosocial) functioning. The higher the score, the more problems the respondent associates with the prompt/sub domain.
Time Frame: At Baseline phone visit
Population: Of the 38 participants assigned to BRITEPath, 28 completed the PedsQOL questionnaire at the baseline timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 28 | 5
score on a scale | 63.1 (12.2) | 70.9 (18.4)

8. Primary Outcome: Quality of Life and Social/Emotional Functioning
Description: as for outcome 7
Time Frame: At 4 week follow up after Baseline
Population: Of the 38 participants assigned to BRITEPath, 25 completed the PedsQOL questionnaire at the 4 week follow-up timepoint. Of the 5 participants assigned to TAU, 4 completed the PedsQOL questionnaire at the 4 week follow-up timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 25 | 4
score on a scale | 71 (11.8) | 64.8 (12)

9. Primary Outcome: Quality of Life and Social/Emotional Functioning
Description: as for outcome 7
Time Frame: At 12 week follow up after Baseline
Population: Of the 38 participants assigned to BRITEPath, 25 completed the PedsQOL questionnaire at the 12 week follow-up timepoint. Of the 5 participants assigned to TAU, 4 completed the PedsQOL questionnaire at the 12 week follow-up timepoint.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 25 | 4
score on a scale | 72.6 (11.5) | 65.5 (13)

10. Secondary Outcome: Application Utilization
Description: Use of the technical components of the BRITEApp for adolescents and young adults will be monitored throughout Phase 1b. Utilization will be measured by the number of participants who have engaged with the application over time, including rating distress levels in the app and utilizing the following app features: learn to savor, reaching out to contacts, soothe breathe, sooth guided meditation, crisis survival strategies, distract with happy thoughts, distract exercise, savor, and soothe activities to help you sleep.
Time Frame: Up to 12 week follow-up
Population: Only 35 of the 38 participants who engaged with the BRITEPath intervention completed baseline and follow up data collection.
  Inconsistency in analyses related to only 35 of 38 participants engaging in the BRITEPath intervention is due to the initial 3 who did not COMPLETE baseline data, but completed a couple demographic questions so they were retained as we intended to treat them.
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 38
Participants
  First distress level: Completed | 24
  First distress level: Did not complete | 14
  Second distress level: Completed | 17
  Second distress level: Did not complete | 21
  Learn to savor: Completed | 2
  Learn to savor: Did not complete | 36
  Reaching out to contacts: Completed | 9
  Reaching out to contacts: Did not complete | 29
  Soothe breathe: Completed | 8
  Soothe breathe: Did not complete | 30
  Soothe guided meditation: Completed | 6
  Soothe guided meditation: Did not complete | 32
  Crisis survival strategies: Completed | 9
  Crisis survival strategies: Did not complete | 29
  Distract with happy thoughts: Completed | 8
  Distract with happy thoughts: Did not complete | 30
  Distract exercise: Completed | 4
  Distract exercise: Did not complete | 34
  Savor: Completed | 5
  Savor: Did not complete | 33
  Soothe activities to help you sleep: Completed | 3
  Soothe activities to help you sleep: Did not complete | 35

11. Secondary Outcome: Application Utilization
Description: Use of the technical components of Guide2BRITE and the BRITEPortal for physicians will be monitored throughout Phase 1b. Utilization will be measured by the number of providers who have completed the Guide2BRITE onboarding process which includes steps 1, 1.2, 1.3, 2, 2.1, 2.2, 2.3, 2.4, 2.5, 3, 3.2, 4, 4.1, and 5.
Time Frame: Up to 12 week follow-up
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 38
Participants
  Step 1: Completed | 28
  Step 1: Did not complete | 10
  Step 1.2: Completed | 28
  Step 1.2: Did not complete | 10
  Step 1.3: Completed | 34
  Step 1.3: Did not complete | 4
  Step 2: Completed | 38
  Step 2: Did not complete | 0
  Step 2.1: Completed | 34
  Step 2.1: Did not complete | 4
  Step 2.2: Completed | 34
  Step 2.2: Did not complete | 4
  Step 2.3: Completed | 34
  Step 2.3: Did not complete | 4
  Step 2.4: Completed | 34
  Step 2.4: Did not complete | 4
  Step 2.5: Completed | 34
  Step 2.5: Did not complete | 4
  Step 3: Completed | 33
  Step 3: Did not complete | 5
  Step 3.2: Completed | 32
  Step 3.2: Did not complete | 6
  Step 4: Completed | 38
  Step 4: Did not complete | 0
  Step 4.1: Completed | 31
  Step 4.1: Did not complete | 7
  Step 5: Completed | 15
  Step 5: Did not complete | 23

12. Secondary Outcome: Service Utilization (Outpatient, School, ER, Legal, Inpatient, Medication) - BRITEPath vs. Treatment as Usual (TAU) at Baseline
Description: The Child and Adolescent Service Assessment (CASA) will collect service utilization of all participants to determine the amount of services accessed in each treatment arm. An overall average of the cost of implementing the BRITEPath intervention (including labor, equipment, supplies, facilitates) will be estimated and between the intervention costs and cost of services used from CASA, a comparison will be made and results published. The CASA response data displayed are those who responded positively that they received the service.
Time Frame: At Baseline phone visit
Population: 33 of 38 participants in BRITEPath intervention and 4 of the 5 TAU participants answered CASA questions.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment As Usual: Participants in the TAU group will not receive the Brite emotion regulation/safety planning app. If participants in the TAU group are determined to be at risk for suicidal ideation or behavior, usual care of a paper-based safety plan will be utilized.
Arm/Group | BRITEPath | Treatment As Usual
Number analyzed (Participants) | 33 | 4
Participants
  Use outpatient services | 32 | 4
  Use school services | 18 | 4
  Use ER services | 12 | 0
  Use legal services | 0 | 0
  Use inpatient services | 8 | 0
  Use medications | 31 | 2

13. Secondary Outcome: Service Utilization (Outpatient, School, ER, Legal, Inpatient, Medication) - BRITEPath vs. Treatment as Usual (TAU) at 4 Week Follow Up
Description: as for outcome 12
Time Frame: At 4 week follow up after Baseline
Population: 32 of 38 participants in the BRITEPath intervention and 4 of the 5 participants in the Treatment As Usual arm of the study responded to CASA questions.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Count of Participants; unit: Participants
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 32 | 4
Participants
  Use outpatient services | 31 | 4
  Use school services | 19 | 4
  Use ER services | 12 | 0
  Use legal services | 0 | 0
  Use inpatient services | 8 | 0
  Use medications | 31 | 2

14. Secondary Outcome: Service Utilization (Outpatient, School, ER, Legal, Inpatient, Medication) - BRITEPath vs. Treatment as Usual (TAU) at 12 Week Follow Up
Description: as for outcome 12
Time Frame: At 12 week follow up after Baseline
Population: 32 of 38 BRITEPath intervention participants and 4 of 5 Treatment As Usual participants completed CASA questions.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Count of Participants; unit: Participants
Arm/Group | BritePath | Treatment As Usual (TAU)
Number analyzed (Participants) | 32 | 4
Participants
  Use outpatient services | 29 | 2
  Use school services | 4 | 0
  Use ER services | 0 | 0
  Use legal services | 0 | 0
  Use inpatient services | 1 | 0
  Use medications | 26 | 2

15. Secondary Outcome: Usability and Satisfaction
Description: Satisfaction to BRITEPath will be assessed through questions developed by investigators to understand experience with the program. Questions investigators have adapted from literature reviews on satisfaction include:
  "If a friend were in need of mental health care for depression or suicidal thoughts or behaviors, would you recommend BRITEPath to help him/her manage symptoms? with answer options of: No, definitely not; No, I don't think so; Yes, I think so; Yes, definitely
  How satisfied are you with the amount of help you received? with answer options of: Dissatisfied; Satisfied; Very Satisfied
  Have the services you received helped you to deal more effectively with your problems? with answer options of: Really didn't help; Yes, somewhat; Yes, a great deal.
Time Frame: At exit interview following week 4 study visit or week 12 study visit (depending on when youth attends mental health session that uses BRITEPath tools)
Population: Out of the 38 participants randomized to receive the BRITE App, only 26 completed the exit interview.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Count of Participants; unit: Participants
Arm/Group | BRITEPath
Number analyzed (Participants) | 26
Participants
  If a friend were in need of mental health care, would you recommend BRITEPath?: No, I don't think so | 3
  If a friend were in need of mental health care, would you recommend BRITEPath?: Yes, I think so | 14
  If a friend were in need of mental health care, would you recommend BRITEPath?: Yes, definitely | 9
  If a friend were in need of mental health care, would you recommend BRITEPath?: Dissatisfied | 0
  If a friend were in need of mental health care, would you recommend BRITEPath?: Satisfied | 0
  If a friend were in need of mental health care, would you recommend BRITEPath?: Very Satisfied | 0
  If a friend were in need of mental health care, would you recommend BRITEPath?: Really didn't help | 0
  If a friend were in need of mental health care, would you recommend BRITEPath?: Yes, somewhat | 0
  If a friend were in need of mental health care, would you recommend BRITEPath?: Yes, a great deal | 0
  How satisfied were you with the amount of help you received?: No, I don't think so | 0
  How satisfied were you with the amount of help you received?: Yes, I think so | 0
  How satisfied were you with the amount of help you received?: Yes, definitely | 0
  How satisfied were you with the amount of help you received?: Dissatisfied | 1
  How satisfied were you with the amount of help you received?: Satisfied | 18
  How satisfied were you with the amount of help you received?: Very Satisfied | 7
  How satisfied were you with the amount of help you received?: Really didn't help | 0
  How satisfied were you with the amount of help you received?: Yes, somewhat | 0
  How satisfied were you with the amount of help you received?: Yes, a great deal | 0
  Have the services you received help you to deal more effectively with your problem?: No, I don't think so | 0
  Have the services you received help you to deal more effectively with your problem?: Yes, I think so | 0
  Have the services you received help you to deal more effectively with your problem?: Yes, definitely | 0
  Have the services you received help you to deal more effectively with your problem?: Dissatisfied | 0
  Have the services you received help you to deal more effectively with your problem?: Satisfied | 0
  Have the services you received help you to deal more effectively with your problem?: Very Satisfied | 0
  Have the services you received help you to deal more effectively with your problem?: Really didn't help | 2
  Have the services you received help you to deal more effectively with your problem?: Yes, somewhat | 20
  Have the services you received help you to deal more effectively with your problem?: Yes, a great deal | 4

16. Secondary Outcome: Usability and Satisfaction
Description: Satisfaction with the technical components of interventions will be assessed through the certain questions from the Post System Satisfaction and Usability Questionnaire (PSSUQ). The PSSUQ is 19 items with response options ranging from 1 to 7 where 1=strongly disagree and 7=strongly agree. The PSSUQ has sub-scores derived from subsets of the questions which reflect system usefulness, information quality, and interface quality. Questions from sub-domains were chosen to tailor the questioning to this particular intervention.
Time Frame: as for outcome 15
Population: Out of the 38 participants randomized to receive the BRITE App, 26 completed the exit interview.
  3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRITEPath
Number analyzed (Participants) | 26
score on a scale
  Overall, I am satisfied with how easy it is to use the BRITE app | 5.7 (1.4)
  The information provided with the BRITE app was clear: number analyzed (Participants) | 25
  The information provided with the BRITE app was clear | 6.2 (1.2)
  The information provided in the BRITE app such as notifications to rate my mood was clear: number analyzed (Participants) | 25
  The information provided in the BRITE app such as notifications to rate my mood was clear | 6.1 (1)
  The information provided during the onboarding with my therapist was clear | 6.5 (0.8)
  I liked interacting with the BRITE app program | 5.8 (1)
  I needed to learn a lot of things before I could get going with the BRITE app | 1.8 (1.2)

17. Secondary Outcome: Cost Estimate for Implementation of BRITEPath Intervention
Description: An overall average of the cost of implementing the BRITEPath intervention (including labor, equipment, supplies, facilitates) will be estimated. Outcome measure data below highlights the estimated cost of the intervention BRITEPath Intervention per participant, measures were based on estimates from staff and not on empirical data at the individual level.
Time Frame: At 12 week follow up after Baseline
Population: 32 of 38 BRITEPath intervention participants interacted with the app. 3 individuals randomized to BRITEPath completed a few demographic questions and were retained as we intended to treat them in the sample. The below measures are based on estimates from staff and not on empirical data at the individual level.
Measure: Mean (Full Range); unit: dollars per participant
Groups:
- BRITEPath Intervention: Participants in the BritePath intervention group receive and emotion regulation/safety planning app.
Arm/Group | BRITEPath Intervention
Number analyzed (Participants) | 32
dollars per participant | 457.43 [214.10 to 597.05]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events at each timepoint (baseline, 4 week follow-up, 12 week follow-up).
Arm/Group | BritePath | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/5
Other Adverse Events (participants affected / at risk) | 0/35 | 0/5

LIMITATIONS AND CAVEATS:
The small sample size of this pilot study was selected for feasibility testing, not for hypothesis testing; thus, inferential tests were underpowered and conducted for exploratory purposes. It lacked a full control group we originally intended to collect, which limits our ability to know whether treatment improvements were due to BRITEPath or to standard care. The impact of treatment on individuals who dropped out of treatment and on those lost during follow-up is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT04000399/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT04000399/ICF_001.pdf